CLINICAL TRIAL: NCT03526393
Title: Construction of the Training Mode Adjustable Equipment Sitting Volleyball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Silvia Regina M. S. Boschi, Principal Investigator, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAEE: 45887715.3.0000.5497
Record Dates: First submitted 2018-04-28; First posted 2018-05-16 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Support Equipment (Experimental): Were selected high performance athletes with various kinds of disabilities found in sitting volleyball functional classification. Three equipment was built to aid high-performance athletes. All the volunteers tested the survey training equipment, attack and serve training equipment and pass training equipment The motor sign captured footage of each athlete, lasted 30 minutes and the data collected provided the data for the construction of the equipment, later there was the interaction of the athletes with the equipment ready to test effectiveness.
  Interventions: Device: Survey training equipment; Device: Attack and serve training equipment; Device: Pass training equipment

INTERVENTIONS:
Device: Survey training equipment — The survey was checking the equipment designed to assist the lifter training survey with greater precision, in aspects of average height of contact of the ball by striker and maximum perimeter of contact with the ball, for the execution of the attack.
Device: Attack and serve training equipment — The attack and serve training equipment was designed to assist the athlete in their body positioning for the execution of the fundamentals of the attack and serve, and the correct extension execution of the of trunk, upper limbs and reaction time of contact with the ball.
Device: Pass training equipment — The equipment for the training of the pass, it was designed to represent the serve forced and technical, variables height, circumference and average speed of the ball. This equipment has been adapted from the conventional volleyball serve equipment, respecting the limits of the sitting volleyball court.

SUMMARY:
The individual adapted sport modalities concentrate most of the technological development for equipment and auxiliary devices, the collective modalities need implements that aid in the development of training and the game.

DETAILED DESCRIPTION:
The individual adapted sport modalities concentrate most of the technological development for equipment and auxiliary devices, the collective modalities need implements that support, in the development of training and the game. It was developed equipment to assist in the training of technical fundamentals and to improve the efficiency of the motor gesture required for the practice of sitting volleyball in athletes with physical disabilities. Ten athletes, sitting volleyball players, were selected to perform a set of technical fundamentals and their variations. Lift the ball (with two variations), attack and serve, and reception. After the analysis of the movements the equipment was elaborated and constructed based on the measurements made with the athletes, such as contact height with the ball, perimeter, speed and parabola.

ELIGIBILITY:
Inclusion Criteria:

* Have functional classification in national or international level,
* Practice experience of sitting volleyball mode of at least five years
* Participate in weekly training at least three times a week.

Exclusion Criteria:

* Non-acceptance of the athlete to participate in the survey
* Does not have the functional classification for the practice of sport

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08-16 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
Ball lifting | 10 minutes
  The survey training equipment helps the athlete to train precision of gesture engine to the trajectory of the ball is more effective and can get in the best conditions to the attacker. 150 repetitions were performed, with 15 seconds interval between tests. Unit of measurement: meter (m) and centimeter (cm)

SECONDARY OUTCOMES:
Attack and loot | 10 minutes
  Equipment for training and assists the athlete on the body positioning during the maximal extension from the execution the fundamentals, for the most suitable length of the trunk and upper limbs. 150 repetitions were made to attack and plunder with 15 seconds interval between tests. Unit of measurement: meter (m) and centimeter (cm).
Pass training | 15 minutes
  The equipment for training the pass was constructed to perform the trajectory of the ball with respect to height, speed and parabola. 150 repetitions were performed for the equipment, with 15 seconds interval between tests. Unit of measurement: kilometers per hour (km/h).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Boschi, PhD, Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Silvia Regina Matos da Silva Boschi, Mogi das Cruzes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No